CLINICAL TRIAL: NCT06611449
Title: The Effect of Minimal Flow Anesthesia on Oxidative and Neuroendocrine Stress Response
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Hilal Deniz, Dr, Resident Doctor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: hdeniz.001
Record Dates: First submitted 2024-05-30; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Low Flow Anesthesia; Oxidative Stress; Neuroinflammatory Response
Keywords: Low Flow Anesthesia; Oxidative Stress; Neuroinflammatory Response

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The minimal flow group (Active Comparator): As soon as mechanical ventilation begins, sevoflurane at a concentration of 3% and a fresh gas flow of 4 L/min with 40-45% oxygen will be used to maintain ventilation until the MAC value reaches 0.9-1.0 For patients in Group 1:the minimal flow group (n=16), maintenance anesthesia will be provided with 80-100% O2 and 3.5-4.5% sevoflurane at a fresh gas flow rate of 0.3-0.5 L/min(minimal fresh gas flow anesthesia) Near the end of the operation, the maintenance anesthetics will be discontinued, and the fresh gas flow will be increased to 6 L/min
  Interventions: Other: The minimal flow anesthesia with sevoflurane group
- The high flow group (Active Comparator): As soon as mechanical ventilation begins, sevoflurane at a concentration of 3% and a fresh gas flow of 4 L/min with 40-45% oxygen will be used to maintain ventilation until the MAC value reaches 0.9-1.0 For patients in Group 2: the high flow group (n=16), maintenance anesthesia will be provided with a 40-45% oxygen-air mixture, 2-2,5% sevoflurane, and a fresh gas flow rate of 4 L/min (high fresh gas flow anesthesia) Near the end of the operation, the maintenance anesthetics will be discontinued, and the fresh gas flow will be increased to 6 L/min
  Interventions: Other: The high flow anesthesia with sevoflurane group

INTERVENTIONS:
Other: The minimal flow anesthesia with sevoflurane group — In the minimal flow group, anesthesia will be maintained with minimal fresh gas flow (0.3-0.5 L/min). The effect of minimal flow anesthesia on oxidative and neuroendocrine stress response will be evaluated by the levels of: IL-6 (proinflammatory cytokine), ACTH (adrenocorticotropic hormone), Cortisol, TAS/TOS (total antioxidant/oxidant status) measured from blood samples.
  Blood samples will be taken from the antecubital area before the surgery begins, thus eliminating the need for repeated invasive procedures. Blood samples will be taken from the patients just before the surgery begins, at the end of the surgery, and at the 6th and 18th hours after the surgery.
  Arms: The minimal flow group
Other: The high flow anesthesia with sevoflurane group — Maintenance of anesthesia in the high flow group will be provided with a high fresh gas flow (4 L/min). The effect of high flow anesthesia on oxidative and neuroendocrine stress response will be evaluated by the levels of: IL-6 (proinflammatory cytokine), ACTH (adrenocorticotropic hormone), Cortisol, TAS/TOS (total antioxidant/oxidant status) measured from blood samples.
  Blood samples will be taken from the antecubital area before the surgery begins, thus eliminating the need for repeated invasive procedures. Blood samples will be taken from the patients just before the surgery begins, at the end of the surgery, and at the 6th and 18th hours after the surgery.
  Arms: The high flow group

SUMMARY:
Patients under general anesthesia who are unconscious and have stopped spontaneous breathing are actively ventilated with anesthesia machines, ensuring the anesthesia gas reaches the lungs and then the bloodstream. Not all the gas reaching the lungs during respiration is used; a small portion is absorbed by the body, and most of it is expelled during exhalation. After eliminating the carbon dioxide in the expired gas, it is more suitable to re-breathe the remaining gas. The portion taken by the patient needs to be provided for the next breath, and this added gas is called "fresh gas flow." Today, low flow anesthesia is defined when the fresh gas flow rate is 0.5-1 L/min, minimal flow anesthesia when it is 0.25-0.5 L/min, and metabolic flow anesthesia when it is 0.25 L/min. Our study will evaluate the effects of minimal flow anesthesia, which is widely used today due to its advantages, on oxidative stress and neuroendocrine stress response

DETAILED DESCRIPTION:
General anesthesia is characterized by anesthesia, analgesia, amnesia, and muscle relaxation. The most common practice today for maintaining anesthesia after induction is to add a low-density effective inhalation anesthetic to an oxygen/air mixture. Patients who are unconscious and have stopped spontaneous breathing are actively ventilated with anesthesia machines, ensuring the anesthesia gas reaches the lungs and then the bloodstream. Minute ventilation refers to the total amount of gas (oxygen, air, and anesthetic agent mixture) a patient breathes in one minute, which is approximately 5-6 L in a normal adult weighing 70 kg.

During respiration, not all the gas reaching the lungs is used; a small portion is absorbed by the body, and most of it is expelled during exhalation. After eliminating the carbon dioxide in the expired gas, it is more suitable to re-breathe the remaining gas for lung physiology, environmental protection, and cost-effectiveness. The portion taken by the patient needs to be provided for the next breath, and this added gas is called "fresh gas flow."

Today, in adults, low flow anesthesia is defined when the fresh gas flow rate is 0.5-1 L/min, minimal flow anesthesia when it is 0.25-0.5 L/min, and metabolic flow anesthesia when it is 0.25 L/min. Reducing the fresh gas flow has positive effects on the patient's health under anesthesia, environmental protection, and cost-effectiveness, as well as reducing pathologies in the operating room staff due to air pollution. Low flow anesthesia has been shown to have no adverse effects on oxygenation, ventilation, organ functions, or hemodynamic parameters. It does not affect any surgical procedure.

The acute stress response associated with surgery and anesthesia is connected to the neuroendocrine-metabolic system and the inflammatory-immune system. In response to surgical stress, adrenocorticotropic hormone(ACTH) is released from the pituitary gland via corticotropin-releasing hormone(CRH). ACTH stimulates the adrenal cortex to release glucocorticoid (cortisol). Both innate and adaptive immune cells play a role in the stress response to surgery. Cytokines mediate the local inflammatory response seen with tissue damage. Pro-inflammatory cytokines, such as interleukin-6 (IL-6), are released, peaking in the first 24 hours post-surgery.

Previous studies have shown an increase in cortisol, ACTH, and IL-6 values on the first postoperative day; their changes were recorded by measuring them at induction, the end of surgery, and at postoperative 12 and 24 hours. The body contains unstable molecules defined as free oxygen radicals. These molecules are balanced by antioxidant molecules. The imbalance in favor of oxidants leads to oxidative stress, causing a series of tissue damage. The biochemical markers indicating this balance are total antioxidant status (TAS) and total oxidative status (TOS).

Our study will evaluate the effects of minimal flow anesthesia, which is widely used today due to its advantages, on oxidative stress and neuroendocrine stress response.

*Research Methodology* Our research is a prospective, randomized controlled clinical study. Patients aged 18-65 undergoing elective septorhinoplasty classified as American Society of Anesthesiologists(ASA) 1-2 will be included. Informed consent will be obtained from patients who volunteer for the study.

Patients included in the study will be divided into two groups using a closed envelope method. After reaching a minimum alveolar concentration (MAC) value of 0.9-1.0, group 1 (minimal flow group) (n=16) will receive maintenance anesthesia with minimal fresh gas flow, and group 2 (high flow group) (n=16) will receive maintenance anesthesia with high fresh gas flow. Group 1 will receive maintenance anesthesia with 80-100% O2 and 3.5-4.5% sevoflurane at a fresh gas flow rate of 0.3-0.4 L/min. Group 2 will receive maintenance anesthesia with 40-45% oxygen-air mixture, 2-2.5% sevoflurane, and a fresh gas flow rate of 4 L/min.

Levels of Total Antioxidant Status (TAS), Total Oxidative Status (TOS), ACTH (adrenocorticotropic hormone), cortisol, and IL-6 (inflammatory cytokine) will be measured from blood samples taken from the patients. Before the surgery, a 20-gauge venous cannula will be placed in the antecubital region for blood sampling to avoid repeated invasive procedures. Immediately before the surgery, 8 ml of blood will be taken as the first sample. The sample will be placed in 3 ml ethylenediaminetetraacetic acid (EDTA) and 5 ml gel tubes and sent to the biochemistry laboratory to be stored at -80°C. At the end of surgery, 5 ml of blood will be taken as the second sample before extubation, placed in a gel tube, and sent to the biochemistry laboratory to be stored at -80°C. At the 6th postoperative hour, 8 ml of blood will be taken as the third sample, placed in 3 ml EDTA and 5 ml gel tubes, and sent to the biochemistry laboratory to be stored at -80°C. At the 18th postoperative hour, 8 ml of blood will be taken as the fourth sample, placed in 3 ml EDTA and 5 ml gel tubes, and sent to the biochemistry laboratory to be stored at -80°C. A total of 30 ml of blood samples will be collected from the patient. The blood samples will be centrifuged at 3000 rpm for 10 minutes, and the separated sera will be stored at -80°C for analysis.

Patients will be discharged with appropriate treatment deemed suitable by the surgical team. The levels of Total Oxidative Status (TOS), Total Antioxidant Status (TAS), ACTH (adrenocorticotropic hormone), cortisol, and IL-6 (inflammatory cytokine) will be measured in the blood sample taken before induction. TAS/TOS will be measured in the second blood sample taken at the end of the surgery. Total Oxidative Status (TOS), Total Antioxidant Status (TAS), ACTH (adrenocorticotropic hormone), cortisol, and IL-6 (inflammatory cytokine) will be measured in blood samples taken at the 6th and 18th postoperative hours. Hemodynamic parameters, visual analogue pain score (VAS), and nausea-vomiting status will be recorded at the 6th and 18th postoperative hours. After centrifuging the blood samples, they will be stored at -80°C, and the specified biomarkers will be evaluated in the laboratory after all samples are collected. The results will be used in our research after statistical analysis.

Data will be analyzed using the Statistical Package for the Social Sciences(SPSS)-statistics 22.0 software package. Categorical variables will be expressed as numbers and percentages, while continuous variables will be presented as median, mean, and standard deviation. The chi-square test will be used to compare differences between categorical variables. The normal distribution of continuous variables will be assessed by the Shapiro-Wilk test. The Student's t-test will be used for parametric data and the Mann-Whitney U test for non-parametric data to compare continuous variables between the two groups. A p-value of <0.05 will be considered significant in all tests.

ELIGIBILITY:
Inclusion Criteria:

* • Ages 18-65

  * Scheduled for elective septorhinoplasty
  * ASA (physical status) 1-2

Exclusion Criteria:

* • ASA (physical status) III-IV

  * Under 18 or over 65
  * Pregnant individuals
  * Serious cardiovascular disease or arrhythmia
  * Chronic obstructive pulmonary disease
  * Severe respiratory failure
  * Uncontrolled cerebrovascular disease
  * Hepatic or renal dysfunction
  * Allergy to propofol, fentanyl, rocuronium, sevoflurane
  * Pituitary gland disease (e.g., pituitary adenoma)
  * Adrenal gland disease (e.g., pheochromocytoma, Cushing's disease)
  * Immune deficiency
  * Neuroendocrine system disease
  * BMI > 40
  * Patients who refuse to provide written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Interleukin 6 (IL-6) level | Just before surgery begins, postoperative 6th hour and postoperative 18th hour
  Proinflammatory cytokines (Biochemical marker)
Adrenocorticotropic hormone (ACTH) level | Just before surgery begins, postoperative 6th hour and postoperative 18th hour
  Adrenocorticotropic hormone(Biochemical marker)
Cortisol level | Just before surgery begins, postoperative 6th hour and postoperative 18th hour
  Biochemical marker
Total oxidative status (TOS) Level | Just before surgery begins, end of surgery, postoperative 6th hour and postoperative 18th hour
  Total oxidative status; blood biochemical tests are used to calculate oxidative indicators.
Total antioxidative status( TAS) Level | Just before surgery begins, end of surgery, postoperative 6th hour and postoperative 18th hour
  Total antioxidative status; blood biochemical tests are used to calculate oxidative indicators.

SECONDARY OUTCOMES:
amount of bleeding | end of surgery
  Total amount of bleeding at the end of surgery
Amount of volatile anesthetic use | End of anesthesia
  Total amount of volatile anesthetic used at the end of anesthesia
Body temperature change | From the beginning of anesthesia to the 18th postoperative hour
  Body temperature measured from the axillary region
The presence of nausea and vomiting | From the recovery of anesthesia to the 18th postoperative hour
  The presence and frequency of nausea and vomiting
Assessment of pain | From the recovery of anesthesia to the 18th postoperative hour
  The severity of the patient's pain is queried according to the visual pain score. The Visual Analog Scale (VAS) is a subjective measure used to assess the intensity of pain a person is experiencing. It consists of a straight line, usually 10 centimeters long, with one end defined as "no pain" and the other end as "worst imaginable pain." Patients are asked to mark a point on this line. As the numerical value increases from 1 to 10, the intensity of the pain increases.
Adverse events | From the recovery of anesthesia to the 18th postoperative hour
  bronchospasm, hypoxemia, airway edema, hypotension, bradycardia, massive bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Resident Doctor, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cusack B, Buggy DJ. Anaesthesia, analgesia, and the surgical stress response. BJA Educ. 2020 Sep;20(9):321-328. doi: 10.1016/j.bjae.2020.04.006. Epub 2020 Jul 21. No abstract available. PMID 33456967
- [Background] Kasikara H, Dumanli Ozcan AT, Bicer CK, Senat A, Yalcin A, Altin C, Mustafa Aksoy S, But A. The effect of low flow anesthesia with sevoflurane on oxidative status: A prospective, randomized study. Saudi Med J. 2022 Mar;43(3):227-235. doi: 10.15537/smj.2022.43.3.20210876. PMID 35256489